CLINICAL TRIAL: NCT00300859
Title: Brief Intervention to Increase Safety Belt Use Among ED Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CDC-NCIPC-0681; 1R49CE000681-01 (NIH)
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Accidents, Traffic

INTERVENTIONS:
Behavioral: brief motivational intervention

SUMMARY:
DESCRIPTION (adapted from applicant's abstract): Injury control experts suggest that consistent SBU is the most effective means for motorists to reduce1he risk of death or serious injury in a crash. Sadly, the SBU prevalence among Massachusetts' residents is among the lowest in the nation. In accord with Healthy People 2010, Objective 15-19, and the CDC's Injury Research Agenda, the investigator will test the utility of a brief intervention to increase SBU among ED patients with self-reported SBU that IS less than "always". A secondary aim is to determine if the brief intervention is more effective among persons being treated for a motor vehicle crash (MVC)-related injury during a "teachable moment" than other non-injured ED patients receiving the same intervention. The research staff will systematically sample ED patients, screening for SBU among eligible participants during a 3-month period. Upon obtaining verbal consent, researchers will ask participants to complete a self-administered screening form on health and safety issues, including SBU. Patients that screen positive, (i.e., give an answer of less than "always use" safety belts) on a SBU screening question will be asked to participate in an intervention to promote health and safety among ED patients. Participants will be reimbursed for their time, and asked to do the following: to give written informed consent via IRB-approved forms and a HIPAA release form; complete an intake form, and agree to a follow-up phone interview at 3 and 6 months post-enrollment. Participants will be randomized into one of two groups: an Intervention Group that will receive a brief intervention designed to increase SBU, and a Control Group that will receive only standard care. Research staff will contact participants for a follow-up phone survey at 3 and 6 months to test the hypothesis that individuals randomized to the Intervention Group will have a higher self-reported SBU than those in the Control Group that received only standard care. Likewise, for the secondary (exploratory) analysis, the hypothesis is that among those treated for MVC-related trauma--and randomized to the intervention group--will have a higher self-reported SBU than others with non MVC-related trauma due to a greater receptivity to brief intervention techniques during the ED visit (i.e. the "teachable moment").

ELIGIBILITY:
Inclusion Criteria:

* ED patients greater than 18 years old, speak English, normal mental status, can give free and autonomous consent,

Exclusion Criteria:

* patient does not have a telephone or is homeless, altered mental status, is a prisoner, under psychiatric evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-02; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
seat belt use

CONTACTS AND LOCATIONS:
Overall Officials: William Fernandez, MD, Principal Investigator — Boston University School of Medicine Dept. of Emergency Medicine